CLINICAL TRIAL: NCT05189639
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multi-centre, Post Marketing Surveillance (PMS) Study of Mylotarg®
Brief Title: A Study To Learn About the Safety Medicine (Called Mylotarg) In People With Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1761035; NCT05189639 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-12-12; First posted 2022-01-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called Mylotarg) for the potential treatment of acute myeloid leukemia (AML). AML is a disease that affects the body's white blood cells. This study is seeking participants in Korea who:

* Are 18 years of age or older
* Are adults and newly diagnosed with AML
* Currently receive Mylotarg for AML treatment in a hospital
* Are capable of a personally signed and dated informed consent document indicating that the participant (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Participant's health will be closely monitored for any unwanted reactions during Mylotarg treatment. Disease progression will also be monitored. This will help determine if Mylotarg is safe to use and its effect on AML treatment.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, non-interventional, multi-centre, PMS to evaluate safety and effectiveness of Mylotarg® in patients with newly-diagnosed CD33-positive AML. As this is a Non-Interventional Study (NIS) all treatment and monitoring of the patients will be at the discretion of the investigator as part of routine practice. The study can be performed in Korean health care centers where Mylotarg® is prescribed to treat AML after obtaining informed consent from the patients as whole case enrollment method.

This study is conducted to determine any problems or questions associated in regard to the following clauses under general clinical practice after marketing Mylotarg®, in accordance with the "Re-examination Guideline of New Drugs, Etc.":

1. Serious Adverse Event (SAE)/Adverse Drug Reaction (ADR)
2. Unexpected Adverse Event (AE)/Adverse Drug Reaction (ADR) that has not been reflected in the approved drug label.
3. Known Adverse Drug Reaction (ADR)
4. Non-Serious Adverse Drug Reaction (Non-SADR)
5. Other safety and effectiveness information

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients newly diagnosed as CD33-positive AML who have been treated* or are being treated* or determined to be treated with Mylotarg® by the investigator's medical decision under routine clinical practice (*patients that have been treated or are being treated with Mylotarg® will be eligible for inclusion during the whole case enrollment period, 2 years after approval date)
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients to whom Mylotarg® is contraindicated as per the local labeling (Patients with a history of hypersensitivity including anaphylaxis to the active substance in Mylotarg® or to any of its components or to any of the excipient.)
* Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly-diagnosed CD33-positive AML in adults
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) | from initiating administration of first dose to the at least 28 calendar days following the last administration of Mylotarg®
  An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent were events between first dose of infusion up to 2 years, that were absent before treatment or that worsened relative to pretreatment state. Serious infections including sepsis (excluding opportunistic infections and tuberculosis) were the pre-defined TEAE of special Interest for this study. AEs included both serious and non-serious adverse events.

SECONDARY OUTCOMES:
Objective Response Rate - Percentage of Participants With Objective Response | assessed after each cycle (each cycle is 7 days) and all cycles (maximum 3 cycles) are administered
  Percentage of participants with OR based assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed remission are those with repeat bone marrow showing less than 5 percent (%) myeloblasts with normal maturation of all cell lines and absolute values of the peripheral blood lasting at least 2 months. PR are those with all CR criteria except at least 50% decrease in the blasts over the pretreatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Seoul national university hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1761035